CLINICAL TRIAL: NCT07002047
Title: Real World and Epidemiology Study of Medically Attended Chlamydia Trachomatis Among Adults in Germany
Status: Active, not recruiting | Type: Observational
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: VAV00049; U1111-1320-4648 (Other: WHO ICTRP)
Record Dates: First submitted 2025-05-23; First posted 2025-06-03 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Chlamydia Trachomatis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Male and Female Adolescents and Adults with CT: Male and Female patients aged between 14 and 44 years of age with documented (confirmed) CT diagnosis

SUMMARY:
This study assesses the epidemiologic situation of chlamydia trachomatis, its complications and long term sequalae and related healthcare resource utilization and costs among adults in Germany.

The study is a retrospective cohort study based on German Statutory Health Insurance (SHI) claims data for adolescents and adults aged 14 to 44 years in the years 2008-2022 with documented (confirmed) diagnosis of CT.

Study Objectives are to:

1. Estimate frequency of potential short-term complications and long-term sequelae in patients with medically attended chlamydia infection
2. Analyze time from first documented prevalent CT infection to first potential complication/sequelae diagnosis
3. Estimate frequency of re-infection (chlamydia recurrence) and co-infections with other sexually transmitted infections (STIs) in patients with medically-attended chlamydia infection
4. Estimate absolute healthcare resource utilization (by level of care and specialty) and costs in patients with chlamydia infection, including for potential short-term complications and long-term sequelae
5. Estimate administrative prevalence of medically-attended chlamydia infection in the overall study population
6. Estimate administrative prevalence of diagnoses potentially associated with a chlamydia infection (i.e., short-term complications/long-term sequelae) in the overall study population
7. Estimate frequency of chlamydia testing in the overall study population

ELIGIBILITY:
Inclusion Criteria:

* Either male or female is documented as gender in base data
* At cohort entry, a patient must be aged between 14 and 44 years

Exclusion Criteria:

* None

Ages: 14 Years to 44 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Adolescents and adults aged 14 to 44 years in the years 2008-2022 with documented (confirmed) diagnosis of CT.
Sampling Method: Non-Probability Sample
Enrollment: 81239 (Actual)
Dates: Start 2025-03-13 (Actual); Primary Completion 2026-02-17 (Estimated); Study Completion 2026-02-17 (Estimated)

PRIMARY OUTCOMES:
Number of female participants with documented (confirmed) outpatient or any inpatient of pelvic inflammatory disease (PID) | From Year 2008 to Year 2022
  The absolute frequency of documented cases will be reported. The relative frequency will be computed as the proportion of patients under exposure (first documented prevalent CT infection) which become cases
Number of female participants with documented confirmed outpatient or any inpatient diagnosis of ectopic pregnancy | From Year 2008 to Year 2022
  The absolute frequency of documented cases will be reported. The relative frequency will be computed as the proportion of patients under exposure (first documented prevalent CT infection) which become cases
Number of female participants with documented confirmed outpatient or any inpatient diagnosis tubal factor infertility | From Year 2008 to Year 2022
  The absolute frequency of documented cases will be reported. The relative frequency will be computed as the proportion of patients under exposure (first documented prevalent CT infection) which become cases
Number of male participants with documented confirmed outpatient or any inpatient diagnosis of orchitis or epididymitis | From Year 2008 to Year 2022
  The absolute frequency of documented cases will be reported. The relative frequency will be computed as the proportion of patients under exposure (first documented prevalent CT infection) which become cases
Number of male participants with documented confirmed outpatient or any inpatient diagnosis of proctitis | From Year 2008 to Year 2022
  The absolute frequency of documented cases will be reported. The relative frequency will be computed as the proportion of patients under exposure (first documented prevalent CT infection) which become cases
Number of male participants with documented confirmed outpatient or any inpatient diagnosis of prostatitis | From Year 2008 to Year 2022
  The absolute frequency of documented cases will be reported. The relative frequency will be computed as the proportion of patients under exposure (first documented prevalent CT infection) which become cases
Number of male and female participants with documented confirmed outpatient or any inpatient diagnosis of female/male infertility | From Year 2008 to Year 2022
  The absolute frequency of documented cases will be reported. The relative frequency will be computed as the proportion of patients under exposure (first documented prevalent CT infection) which become cases
Number of male and female participants with documented confirmed outpatient or any inpatient diagnosis of Urethritis and urethral syndrome | From Year 2008 to Year 2022
  The absolute frequency of documented cases will be reported. The relative frequency will be computed as the proportion of patients under exposure (first documented prevalent CT infection) which become cases
Time in days from first documented prevalent CT infection to first documented complication/sequelae diagnosis | From Year 2008 to Year 2022
  This time-to-event analysis will use the Kaplan-Meier method to estimate the median time-to-event in the presence of censoring
Number of male and female participants with confirmed outpatient or any inpatient CT diagnosis at least 30 days after last CT diagnosis of any kind (reinfection) | From Year 2008 to Year 2022
  The absolute number of documented cases will be reported. The relative frequency will be computed as the proportion of patients under exposure (first documented prevalent CT infection) which become cases.
Number of CT reinfections/episodes | From Year 2008 to Year 2022
  The absolute number of documented cases will be reported. The relative frequency will be computed as the proportion of patients under exposure (first documented prevalent CT infection) which become cases.
Number of male and female participants with documented confirmed outpatient or any inpatient diagnosis of other STI | From Year 2008 to Year 2022
  The absolute number of documented cases will be reported. The relative frequency will be computed as the proportion of patients under exposure (first documented prevalent CT infection) which become cases.
Cost incurred from the number of physician contacts (of any specialty) | From Year 2008 to Year 2022
  Costs are summed up per patient for the specified follow-up time
Costs incurred from the number of hospital admissions | From Year 2008 to Year 2022
  Costs are summed up per patient for the specified follow-up time
Costs incurred for the number of prescriptions filled for any drug | From Year 2008 to Year 2022
  Costs are summed up per patient for the specified follow-up time
Costs incurred for the number of filled prescriptions for any medical aid | From Year 2008 to Year 2022
  Costs are summed up per patient for the specified follow-up time
Costs incurred for the number of physician contacts (of any specialty) related to CT or STI-diagnoses. | From Year 2008 to Year 2022
  Costs are summed up per patient for the specified follow-up time
Costs incurred for the number of hospital admissions related to CT or STI-diagnoses. | From Year 2008 to Year 2022
  Costs are summed up per patient for the specified follow-up time
Costs incurred for the number of filled prescriptions for CT-related antibiotics, dispensed within 30 days after CT diagnosis | From Year 2008 to Year 2022
  Costs are summed up per patient for the specified follow-up time and numbers for each ATC code will be reported separately and in aggregated form
Costs incurred for the number of filled prescriptions for medical aids related to CT or STI diagnoses | From Year 2008 to Year 2022
  Costs are summed up per patient for the specified follow-up time
Total CT-/STI-unspecific health care costs (inpatient, outpatient, drugs, medical aids) | From Year 2008 to Year 2022
  Costs are summed up per patient for the specified follow-up time
CT-/STI-unspecific outpatient costs | From Year 2008 to Year 2022
  Costs are summed up per patient for the specified follow-up time
CT-/STI-unspecific inpatient costs | From Year 2008 to Year 2022
  Costs are summed up per patient for the specified follow-up time
CT-/STI-unspecific drug cost | From Year 2008 to Year 2022
  Costs are summed up per patient for the specified follow-up time
CT-/STI-unspecific medical aid costs | From Year 2008 to Year 2022
  Costs are summed up per patient for the specified follow-up time
Outpatient costs that are related to cases with a confirmed CT diagnosis | From Year 2008 to Year 2022
  Costs are summed up per patient for the specified follow-up time
Inpatient costs that are related to cases with any CT diagnosis | From Year 2008 to Year 2022
  Costs are summed up per patient for the specified follow-up time
Outpatient costs that are related to cases with any confirmed STI diagnosis | From Year 2008 to Year 2022
  Costs are summed up per patient for the specified follow-up time
Inpatient costs that are related to cases with any confirmed STI diagnosis | From Year 2008 to Year 2022
  Costs are summed up per patient for the specified follow-up time
Costs of potentially CT-relevant antibiotics dispensed up to 30 days after confirmend outpatient or any inpatient CT diagnosis | From Year 2008 to Year 2022
  Costs are summed up per patient for the specified follow-up time

SECONDARY OUTCOMES:
Confirmed outpatient or any inpatient CT diagnosis | From Year 2008 to Year 2022
  The absolute number of prevalent cases per calendar year will be reported for each outcome. Due to the possibility of multiple infections per person the number of affected individuals will also be reported. The relative frequency will be computed as the proportion of patients which become cases
Confirmed outpatient or any inpatient of PID (CT associated, or other origin) in females | From Year 2008 to Year 2022
  The absolute number of prevalent cases per calendar year will be reported for each outcome. Due to the possibility of multiple infections per person the number of affected individuals will also be reported. The relative frequency will be computed as the proportion of patients which become cases
First documented confirmed outpatient or any inpatient diagnosis of ectopic pregnancy in females | From Year 2008 to Year 2022
  The absolute number of prevalent cases per calendar year will be reported for each outcome. Due to the possibility of multiple infections per person the number of affected individuals will also be reported. The relative frequency will be computed as the proportion of patients which become cases
First documented confirmed outpatient or any inpatient diagnosis tubal factor infertility in females | From Year 2008 to Year 2022
  The absolute number of prevalent cases per calendar year will be reported for each outcome. Due to the possibility of multiple infections per person the number of affected individuals will also be reported. The relative frequency will be computed as the proportion of patients which become cases
First documented confirmed outpatient or any inpatient diagnosis of orchitis or epididymitis in males | From Year 2008 to Year 2022
  The absolute number of prevalent cases per calendar year will be reported for each outcome. Due to the possibility of multiple infections per person the number of affected individuals will also be reported. The relative frequency will be computed as the proportion of patients which become cases
First documented confirmed outpatient or any inpatient diagnosis of proctitis in males | From Year 2008 to Year 2022
  The absolute number of prevalent cases per calendar year will be reported for each outcome. Due to the possibility of multiple infections per person the number of affected individuals will also be reported. The relative frequency will be computed as the proportion of patients which become cases
First documented confirmed outpatient or any inpatient diagnosis of prostatitis in males | From Year 2008 to Year 2022
  The absolute number of prevalent cases per calendar year will be reported for each outcome. Due to the possibility of multiple infections per person the number of affected individuals will also be reported. The relative frequency will be computed as the proportion of patients which become cases
First documented confirmed outpatient or any inpatient diagnosis of infertility in males | From Year 2008 to Year 2022
  The absolute number of prevalent cases per calendar year will be reported for each outcome. Due to the possibility of multiple infections per person the number of affected individuals will also be reported. The relative frequency will be computed as the proportion of patients which become cases
First documented confirmed outpatient or any inpatient diagnosis of Urethritis and urethral syndrome in males | From Year 2008 to Year 2022
  The absolute number of prevalent cases per calendar year will be reported for each outcome. Due to the possibility of multiple infections per person the number of affected individuals will also be reported. The relative frequency will be computed as the proportion of patients which become cases
Number of male and female participants with documented CT test (screening) | From Year 2008 to Year 2022
  The absolute number of tests as well as the absolute and relative frequency of tested individuals will be reported
Number of male and female participants with documented CT tests (diagnostic/curative) | From Year 2008 to Year 2022
  The absolute number of tests as well as the absolute and relative frequency of tested individuals will be reported

CONTACTS AND LOCATIONS:
Locations (1):
- Germany, Germany

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to the study report and the statistical analysis plan. Access to patient-level data cannot be granted due to data protection regulations applicable to the processing of secondary data for health services research.
  Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org